CLINICAL TRIAL: NCT05315986
Title: The Gut-sleep-brain Axis: Targeting the Gut Microbiota and Sleep Quality by Individualized Non-pharmaceutical Approaches to Promote Healthy Ageing.
Brief Title: Exploration of Relationships Between Sleep, Gut Health and Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: R210281
Record Dates: First submitted 2022-02-21; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Insomnia; Sleep Disturbance
Keywords: sleep; polysomonography; food supplement; gut health; microbiome; cognition; EEG; Dreem3
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Intervention Model Description: Forty-eight (i.e. n=12 per group; 4 groups) healthy older adults aged 55 and over with subjective sleep complaints will be recruited for this 4-week double blinded placebo controlled feasibility study. This project will adopt a 2 x 2 Factorial design.
Who Masked: Participant, Investigator
Masking Description: Participant's and Investigators will be blinded to which participants are receiving the dietary saffron supplement and placebo. Random allocation will be conducted by an independent researcher.
  Participants and investigators will not be blinded to which participants have been allocated ot the ESE intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Sleep intervention (ESE) & Saffron (food supplement) (Experimental): Saffron: Dietary supplement consists of a gummy sweet (Saffr'Inside; 30mg). Ingest one gummy per day for a duration of 4 weeks total.
  Enhanced Sleep Education (ESE): Receive a psycho-education based multi-component sleep intervention consisting of: Sleep education, Sleep hygiene, mindfulness and sleep behavioural recommendations adapted from the validated Brief Behaviour Treatment for Insomnia (BBTi) intervention.The intervention is presented to participants via a pre-recorded presentation, lasting approximately 15 minutes. Participants will also receive some personalized feedback from their objective sleep measurements, collected from their EEG data to help them better understand their sleep patterns.
  Interventions: Dietary Supplement: Saffr'Inside; 30mg; Behavioral: Enhanced Sleep Education
- Group 2: Sleep intervention (ESE) & No Saffron (placebo food supplement) (Experimental): Placebo (no Saffron): Placebo food supplement identical looking (gummy sweet) to experimental food supplement. Ingestion of one gummy per day for a duration of 4 weeks total.
  Enhanced Sleep Education (ESE): Receive a psycho-education based multi-component sleep intervention consisting of: Sleep education, Sleep hygiene, mindfulness and sleep behavioural recommendations adapted from the validated Brief Behaviour Treatment for Insomnia (BBTi) intervention.The intervention is presented to participants via a pre-recorded presentation, lasting approximately 15 minutes. Participants will also receive some personalized feedback from their objective sleep measurements, collected from their EEG data to help them better understand their sleep patterns.
  Interventions: Behavioral: Enhanced Sleep Education; Dietary Supplement: Placebo food supplement
- Group 3: No sleep intervention (Control ESE) & Saffron (food supplement) (Experimental): Saffron: Dietary supplement consists of a gummy sweet (Saffr'Inside; 30mg). Ingest one gummy per day for a duration of 4 weeks total.
  No Psycho-education (ESE) intervention. Control.
  Interventions: Dietary Supplement: Saffr'Inside; 30mg
- Group 4: No sleep intervention (Control ESE) & No Saffron (placebo food supplement) (Placebo Comparator): Placebo (no Saffron): Placebo food supplement identical looking (gummy sweet) to experimental food supplement. Ingestion of one gummy per day for a duration of 4 weeks total.
  No Psycho-education (ESE) intervention. Control.
  Interventions: Dietary Supplement: Placebo food supplement

INTERVENTIONS:
Dietary Supplement: Saffr'Inside; 30mg — Ingestion of one gummy sweet of Saffr'Inside; 30mg, on a daily basis for 4 weeks.
  Arms: Group 1: Sleep intervention (ESE) & Saffron (food supplement); Group 3: No sleep intervention (Control ESE) & Saffron (food supplement)
Behavioral: Enhanced Sleep Education — Psycho-education based multi-component sleep intervention
  Arms: Group 1: Sleep intervention (ESE) & Saffron (food supplement); Group 2: Sleep intervention (ESE) & No Saffron (placebo food supplement)
Dietary Supplement: Placebo food supplement — Placebo food supplement identical to the active gummy sweet of Saffr'Inside; 30mg, on a daily basis for 4 weeks.
  Arms: Group 2: Sleep intervention (ESE) & No Saffron (placebo food supplement); Group 4: No sleep intervention (Control ESE) & No Saffron (placebo food supplement)

SUMMARY:
Our study aims to build on emerging evidence showing relationships between gut health, sleep and brain functions. To achieve this, our study aims to test the feasibility of using non-pharmacological interventions: a psychoeducation-based intervention (enhanced sleep education - ESE) and a dietary supplement (Saffron extract), to improve sleep in older adults with insomnia complaints. Our study also aims to test the feasibility of using wearable and commercially available EEG headband technology to measure objective sleep quality in the home, which will allow for a reliable and ecologically more valid sleep research.

DETAILED DESCRIPTION:
One-third of the UK adult population presents with disordered sleep, and the prevalence further increases with ageing. Disordered sleep has also been identified as a risk factor for dementia, which is alarming given that cases of dementia are predicted to triple across the world by 2050.

Our study aims to build on emerging evidence showing relationships between gut health, sleep, and brain functions. To achieve this, our study aims to test the feasibility of using non-pharmacological interventions: a psychoeducation-based intervention (enhanced sleep education - ESE) and a dietary supplement (Saffron extract), to improve sleep in older adults with insomnia. The study aims to test the feasibility of using wearable sleep tracking EEG technology (DREEM3 device) to measure sleep quality in the home environment, which could contribute to a reliable but naturalistic and accessible future sleep research.

The study is split into 4 phases:

Screening phase: Participants will be asked to complete an online screening assessment to check for eligibility.

Baseline assessment phase (1 week): Participants will complete in-person testing in the Sleep and Brain Research Unit (SBRU) located at the University of East Anglia, to assess their cognitive functions, psychological well-being, and postural control. They will be asked to provide a faecal sample to profile the baseline gut microbiota, a urine sample to gain a baseline measure for testing supplement adherence and wear the DREEM3 headband device and complete a sleep diary to track their sleep quality with a high accuracy in their habitual home environment.

Intervention phase (4 weeks): Participants will be randomly assigned to 1 of 4 groups following a factorial design: Group 1: Food supplement & ESE; Group 2: Food supplement & No ESE (control); Group 3: Placebo (control) & ESE, and Group 4: Placebo (control) & No ESE (control). These groups will allow us to test the effectiveness of each non-pharmacological intervention for feasibility.

Follow-up assessment (1 week - overlap with the last week of intervention): Participants will be asked to measure their sleep at home using the DREEM3 EEG device and complete a sleep diary, and finally will be re-tested for cognitive performance, psychological wellbeing, and postural control. A follow-up faecal sample and urine sample will be collected as well.

This research predicts that it is feasible for sleep difficulties in older adults to be objectively assessed in the home environment and non-pharmacologically treated using food supplements and behavioural techniques. It endeavours to provide pilot evidence for the effectiveness of future individualized non-pharmaceutical sleep treatments in older people at risk of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 55 years
2. Conversational English and capacity to consent
3. Availability to take part in the study
4. Subjective sleep complaints of impaired sleep quality or insufficient sleep
5. Participants with no clinical diagnosis or signs of dementia (m-ACE-III score above 21)
6. Potential for sleep complications such as insomnia before the study
7. A body mass index between 20 and 35 for men, and 18.5 and 35 for women
8. High Score on Pittsburgh Sleep Quality Index (PSQI; > 5) OR The Insomnia Severity Index (ISI; > 10)

Exclusion Criteria:

1. Acute infections or diseases
2. Psychiatric disorders or chronic neurological conditions include a diagnosis of dementia, mild cognitive impairment (MCI)/ prodromal AD.
3. Learning, sensory, or motor impairment/ disabilities that would pose an unfair disadvantage in the cognitive tests
4. Chronic pain conditions
5. Currently taking blood thinning medications
6. Current diagnosis of malignant tumours/ cancers
7. Worked as a shift worker or travelled across more than three time zones in the past two months
8. Alcohol consumption above 14 units/week and/ use or dependency of illicit substances/alcohol
9. Consume more than 5 cups of caffeinated beverages (e.g., coffee/tea/coke, etc) per day.
10. Smokers (tobacco, e-cigarettes, or vapes)
11. Taking antibiotics, or any dietary supplements that may interfere with study outcomes.
12. Self-quarantined or presumed positive status for COVID-19 (see considerations for COVID-19 in safety and comfort section).
13. Currently enrolled or enrolled previously (within the last 2 months) in a drug trial.
14. Participants who show signs or symptoms of having dementia.
15. Participants with high scores (>10) on the Patient Heath Questionnaire-9 (PHQ-9) depression scale and/ or who indicate that they have suicidal thoughts
16. A diagnosis of untreated sleep apnoea or another sleep-related disorder excluding insomnia

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-04-29 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of nights on which participants used the Dreem headband over a 14 day period | 2 weeks
  Frequency of Dreem headband usage over a 14 day period will be used to measure device adherence rates. Higher adherence rates will indicate higher levels of acceptability of the device as a method of measuring electrical activity (electroencephalogram) within the home environment
Mean percentage of Dreem device signal quality over a 14 day period | 2 weeks
  Signal quality will range from 0-100%, with percentages >80% indicating good signal quality. Higher signal quality will indicate higher levels of feasibility of the device as a method of measuring objective sleep quality based on electrical activity of the brain (electroencephalogram) within the home environment.
Number of Participants who report that they made changes to their sleeping habits following engagement in Enhanced Sleep Education (ESE). | 4 weeks
  Frequency of participants who make self-reported changed to their sleeping habits will be used to measure adherence rates to the Enhanced Sleep Education (ESE) intervention. Higher adherence to the intervention will indicate higher acceptability of this method for treating sleep complaints.
Changes in scores on the self-reported sleep quality measure using the Pittsburgh Sleep Quality Index (PSQI) pre/post treatment conditions compared to a placebo. | 4 weeks
  Changes in scores on the Pittsburgh Sleep Quality Index (PSQI) pre/post treatment conditions compared to a placebo will be used to measure feasibility of using proposed treatment conditions to treat sleep difficulties. Treatment conditions include: Enhanced Sleep Education (ESE) intervention X Dietary Supplement (Saffr'Inside), ESE X Placebo, No ESE (control) X Dietary Supplement (Saffr'Inside), No ESE (control) X Placebo. A decrease in scores on the PSQI would indicate improved sleep and suggest feasibility of using the described treatment conditions to improve subjective sleep complaints. (Highest score = 21, Lowest score = 0)
Changes in scores on the Insomnia Severity Index (ISI) pre/post treatment conditions compared to a placebo. | 4 weeks
  Changes in Insomnia Severity Index (ISI) pre/post treatment conditions compared to a placebo will be used to measure feasibility of using proposed treatment conditions to treat sleep difficulties. Treatment conditions include: Enhanced Sleep Education (ESE) intervention X Dietary Supplement (Saffr'Inside), ESE X Placebo, No ESE (control) X Dietary Supplement (Saffr'Inside), No ESE (control) X Placebo. A decrease in scores on the ISI would indicate improved sleep and suggest feasibility of using the proposed treatment conditions to improve subjective sleep complaints. (Highest score = 28, Lowest score= 0)
Changes in objective sleep quality as measured by the sleep efficiency index based on the Dreem electroencephalogram headband pre/post treatment conditions compared to a placebo. | 4 weeks
  Sleep efficiency index will be measured using percentage (sleep efficiency = total sleep time / time in bed x 100).
  Changes in sleep efficiency index of sleep will be used to measure the feasibility of the proposed treatment conditions on improving objective sleep quality. Higher percentages of sleep efficiency suggest improved sleep.
Changes in the time spent awake following initial sleep onset (in minutes) as measured by the Dreem electroencephalogram headband pre/post treatment conditions compared to a placebo. | 4 weeks
  Changes in the time spent awake following initial sleep onset (in minutes) will be used to measure objective sleep quality. Decreases in time spent awake following initial sleep onset (in minutes) will suggest feasibility of proposed treatment conditions for improving objective sleep quality.
Mean number of days on which participants ingested the dietary supplements (Saffr'Inside) per subject over a 4 week period | 4 weeks
  Frequency (mean number of days per subject) of ingestion of the dietary supplement will be used to measure the adherence rate of the supplement. Higher adherence rates will indicate higher levels of acceptability of using a supplement to improve sleep complaints.

SECONDARY OUTCOMES:
Changes in scores on the Patient Health Questionnaire (PHQ-9) pre/post treatment conditions compared to a placebo. | 4 weeks
  Changes in scores on the Patient Health Questionnaire (PHQ-9) pre/post treatment conditions compared to a placebo will be used to measure the feasibility of proposed treatment conditions to improve Psychological wellbeing. A decrease in scores indicates a decrease in experiences of low mood and improved psychological wellbeing. (highest score = 27, lowest score = 0)
Changes in the time to complete (in seconds) on the Trail Making Task B pre/post treatment conditions compared to a placebo. | 4 weeks
  Changes in completion time (in seconds) on the Trail Making Task B pre/post treatment conditions compared to a placebo will be used measure changes in participants cognitive functioning. Decreases in completion time would suggest improve cognitive functioning.

OTHER OUTCOMES:
Changes in gut microbiome composition following a period of ingesting a dietary supplement (Saffr'Inside) | 4 weeks
  To examine species composition, we will perform community analysis via 16S rRNA sequencing. DNA will be extracted from faecal samples and a 250bp region from the V3-V4 hyper-variable region amplified and sequenced on the Illumina MiSeq platform. Principle coordinates analysis (PCoA) of UniFrac/Bray-Curtis distances and ANOSIM/PERMANOVA tests will be used to identify differences in microbial community structure between control and treatment groups pre/post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alpar S Lazar, PhD, Principal Investigator — University of East Anglia

IPD SHARING:
Plan to Share IPD: Yes
IPD may include: Participant contact details, Participant demographic information, Participant scores on screening questionnaires and DNA extracted from urine/fecal samples.
  Data will be shared with other researchers within the University of East Anglia (UEA) if Participants consent to this, so that individuals can be contacted of similar research studies going on at the UEA that they may be eligible to be enrolled in.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available following completion of the study for a minimum of 10 years.
Access Criteria: Data will only be shared with researchers at the UEA.